CLINICAL TRIAL: NCT05890989
Title: Relationship Between Epicardial Adipose Tissue Thickness and Sedentary Time, Physical Activity Level, and Physical Performance in Patients With Hypertension
Brief Title: Relationship of Epicardial Adiposity With Sedentary Time, Physical Activity and Performance in Hypertensives
Status: Completed | Type: Observational
Sponsor: Karamanoğlu Mehmetbey University (Other)
Collaborators: Karaman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Emine Tunç Süygün, LECTURER, Karamanoğlu Mehmetbey University
Other Study IDs: KMU-TUNCSUYGUN-001
Record Dates: First submitted 2023-05-16; First posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Hypertension
Keywords: Epicardial adipose tissue; Hypertension; Physical activity; Sedentary time; Physical performance
MeSH Terms: conditions — Hypertension; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- INCREASED EPICARDIAL ADIPOSIS TISSUE
  Interventions: Diagnostic Test: EPICARDIAL ADIPOSIS TISSUE AND PHYSICAL PERFORMANCE MEASUREMENT

INTERVENTIONS:
Diagnostic Test: EPICARDIAL ADIPOSIS TISSUE AND PHYSICAL PERFORMANCE MEASUREMENT — EPICARDIAL ADIPOSIS TISSUE AND PHYSICAL PERFORMANCE MEASUREMENT OF THE PARTICIPANTS WAS MADE.

SUMMARY:
Epicardial adipose tissue is associated with the development of cardiovascular disease and its increase is positively correlated with blood pressure elevation in hypertensive individuals. In the literature, being physically active has been shown to be effective in the treatment of hypertension and reduction of epicardial adipose tissue thickness. The aim of this study was to evaluate the relationship between epicardial adipose tissue thickness and sedentary time, physical activity level and physical performance in patients with hypertension. The study included 40 patients with hypertension. The physical and demographic characteristics of the participants were collected using a sociodemographic form. Waist/hip circumference was measured with tape measure and epicardial adipose tissue thickness with echocardiography device. Physical activity levels and sedentary time were recorded via IPAQ-7. Physical performance was determined using the 30-s sit-and-stand test. There is no previous study in the literature evaluating the relationship between epicardial adipose tissue thickness and sedentary time and physical activity levels in hypertensive patients. With this study, we aim to contribute to the literature by filling this deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being diagnosed with hypertension for at least 6 months
* Speaking Turkish
* to be able to read and write,
* To be between 18-65 years old

Exclusion Criteria:

* Severe valvular disease
* be heart failure
* being cardiomyopathy
* having chronic kidney disease
* being thyroid diseases
* active infectious or inflammatory diseases
* serious psychiatric illnesses such as panic disorder or major depression

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers who had been diagnosed with hypertension for at least 6 months
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
EPICARDIAL ADIPOSIS TISSUE MEASUREMENT | measured at admission
  All patients underwent transthoracic echocardiography conducted by a single cardiologist using a Philips HD11XE (Philips Medical Systems) device in the left lateral decubitus position by the standard technique. Epicardial fat thickness was measured in the parasternal long axis imaging window, using the aortic annulus as an anatomical indicator for vertical measurement, and the widest part of the region from the right ventricular free wall to the pericardium at the end of the systole.

SECONDARY OUTCOMES:
PHYSICAL PERFORMANCE | measured at admission
  The physical performance of the participants was evaluated with the 30-second sit-and-stand test. While seated in a chair with a seat height of 43.2 cm and a supported back, the patient was asked to stand up and sit down as quickly as possible while crossing his/her hands over his/her chest. The 30-second duration of the test was monitored with a stopwatch and the number of times the participant stood up and sat down was noted. Two trials were performed before the test.

OTHER OUTCOMES:
PHYSICAL ACTIVITY | measured at admission
  Physical activity level was evaluated with the Turkish version of the International Physical Activity Questionnaire-7 (IPAQ-7), whose reliability and validity were confirmed by Saglam et al. The IPAQ-7 is a seven-item questionnaire that assesses severe physical activity (duration: min and frequency: day), moderate physical activity (duration: min and frequency: day), and walking time of at least 10 minutes (frequency: day) over the previous seven days. The metabolic equivalent of task (MET) corresponding to the basal metabolic rate is converted from severe and moderate activity and walking periods, and the overall physical activity score (MET- min/week) is determined
SEDENTARY TIME | measured at admission
  Sedentary time was questioned with the International Physical Activity Questionnaire-7 (IPAQ-7), the reliability and validity of which was confirmed by Saglam et al.

CONTACTS AND LOCATIONS:
Locations (1):
- Karamanoğlu Mehmetbey University, Karaman, Turkey (Türkiye)